CLINICAL TRIAL: NCT06192875
Title: A Novel Molecular Approach to Blood DNA Screening for Cancer: Specificity Assessment (The NOMAD Study)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 15-006191; NCI-2023-09354 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-006191 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — With participant permission, samples will be stored for future research. If future studies examine DNA and findings are noted, the participant will be notified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood and urine sample collection on study. Patients' medical records are reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to establish "normal' values for a new blood test and urine test approach to cancer screening. Patients undergo blood and urine sample collection on study. Patients' medical records are reviewed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess blood level distributions of candidate methylated DNA tumor markers across a cohort of patients without known cancer or precancer and, thereby, to estimate specificity cutoffs across a range of percentiles.

II. To evaluate the effects on marker levels (or test specificity) of selected demographic, exposure, medication, and chronic disease covariates.

III. To build a biospecimen archive to facilitate assessment of clinical specificity in future molecular blood test studies or appraisal of test refinements.

IV. Assess feasibility for detection of cancer using urine samples to assay MDMs, RNA or protein in cell free or extra-cellular vesicles.

V. Assess feasibility for detection of cancer using saliva to assay MDMs, RNA or protein in cell free or extra-cellular vesicles.

ELIGIBILITY:
Inclusion Criteria:

* 10,000 patients without a known internal (non-cutaneous) cancer or a history of an internal cancer

  * To balance age, rough recruitment goals will be set for the following subsets: 18-39 years, 40-49 years , 50-59 years , 60-69 years , 70-79 years , and >= 80 years
  * To balance sex, roughly half of the participants recruited within each age subset will be women
  * Roughly half of all participants will have had a colonoscopy or colon x-ray within the past 5 years, or Cologuard® test in the last 3 years which were negative for cancer and precancerous lesions
  * Roughly half of all participants will have had a chest x-ray within the past 5 years which was negative for cancer
  * Roughly half of women participants will have had a mammography in the past 5 years which was negative for cancer
  * An attempt will be made to recruit minimums (parentheses) of the following subsets: men with normal Prostate-specific antigen (PSA) level (200); diabetes mellitus (200); connective tissue diseases like rheumatoid arthritis, systemic lupus erythematosus, and scleroderma (100); chronic obstructive lung disease (100); inflammatory bowel disease or cirrhosis (100), and pancreatitis (100)
  * To assess the effects of other common covariates, specific recruitment targets will not be set. Rather, data obtained on all participants will include BMI, smoking (past/present), alcohol consumption, pregnant status (women), and selected medications (steroidal and non-steroidal anti-inflammatory drugs, statins, anti-hypertensives, and anti-depressants)

Exclusion Criteria:

* Patients has a past or current diagnosis of invasive cancer (this does not include basal cell or squamous cell skin cancers)
* Patient has had a solid organ transplant
* Inability to give informed consent

URINE EXCLUSIONS

* Patient has transurethral instrumentation (cystoscopy, placement of urinary catheter) within the 7 days prior to sample collection
* Patient has chronic indwelling urinary catheter
* Patient has had a urinary tract infection within the 14 days prior to sample collection

SALIVA EXCLUSIONS

* Patient has known clinically significant xerostomia
* Patient has known recent (within 30 days prior to collection) active upper respiratory tract infection or anogenital infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without a known internal (non-cutaneous) cancer or a history of an internal cancer
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-09-28 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Blood level distributions of methylated DNA tumor markers | Baseline
  Assessed through assays performed on blood plasma across a cohort of patients without known cancer or precancer to estimate specificity cutoff ranges.
Biospecimen archive | Up to study completion (estimate 20 years)
  Assessed by total number of blood samples collected. Collected blood samples will be used to facilitate assessment of clinical specificity in future molecular blood test studies or appraisal of test refinements.
Detection of cancer using urine samples | Baseline
  Assessed by number of urine samples used to assay methylated DNA markers (MDMs), RNA, or protein in cell free or extracellular vesicles.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Kisiel, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials